CLINICAL TRIAL: NCT07159789
Title: Non-Invasive Neuromodulation in MS Induced Spastic Paraparesis
Brief Title: Repetitive Transcranial Magnetic Stimulation (rTMS) in MS Induced Spastic Paraparesis
Acronym: CeV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Neuro-Outaouais (Other)
Collaborators: University of Ottawa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CeV
Record Dates: First submitted 2025-08-29; First posted 2025-09-08 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis
Keywords: rTMS; Neuromodulation; MS Induced Spastic Paraparesis; Spastic paresis; neural synchrony; neuroplasticity
MeSH Terms: conditions — Multiple Sclerosis | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Patient will be randomized in a 1:1 ratio, into two parallel groups. Randomization will be stratified according to age, ongoing use or not of Fampridine and baseline timed 25-foot walk test (T25FWT) results
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rTMS (repetitive Transcranial Magnetic Stimulation ) (Active Comparator): rTMS will use 100% magnetic pulses to stimulate specific areas of the brain
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- sham rTMS (Sham Comparator): Sham rTMS will be conducted using the same DCC coil and MagStim machine but using only 10% of maximum machine output as stimulation intensity
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — Treatment with the rTMS or sham rTMS will be scheduled daily 5x per week for a total of 6 consecutive weeks followed, after a 6 week pause, by another treatment session of 6 weeks where all patients will receive active rTMS treatment

SUMMARY:
Study the impact of rTMS on walking ability in people with Multiple Sclerosis (MS) induced spastic paraparesis and moderate walking disability.

DETAILED DESCRIPTION:
Measure the impact of rTMS on overall disability level, walking endurance, quality of life parameters, and corroborate with EEG parameters of neural synchrony in patients with MS.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Age ≥ 18 years and less than 71 years.
3. Diagnosis of MS according to the revised 2017 McDonald Criteria (Thompson et al. 2018).
4. EDSS of 3.0 to 6.5 with a pyramidal functional system score of 3.0 or more.
5. Neurologically stable with no change in symptom related medications or relapse for at least 30 days prior to screening.
6. Patients will be allowed to continue fampridine provided they started more than 30 days prior to screening. They will not be allowed to start fampridine, any stimulant (modafenil, methylphenidate etc) or symptomatic treatment of spasticity (baclofen, tizanidine, botulinum toxin etc.) during the study.
7. No change in disease modifying therapy for at least 3 months prior to screening.
8. Ability to perform T25FWT, the MSQoL 6MWT Ability and willingness, in the investigator's opinion, to comply with the study protocol.

Exclusion Criteria:

1. Know presence of other neurologic disorders, which in the opinion of the investigator could add to the patient's neurological disability within the timespan of the study.
2. Evidence of clinically significant cardiovascular (including arrhythmias), psychiatric, pulmonary, renal, hepatic, endocrine, metabolic, or gastrointestinal disease that, in the investigator's opinion, would preclude patient participation.
3. Pregnant or breastfeeding or intending to become pregnant during the study.
4. Any previous rTMS therapy for any indication.
5. Presence of any contraindication to rTMS therapy such as but not limited to: CNS implanted devices, pacemaker.
6. Any condition which in the opinion of the investigator will render the patient unsuitable to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Improvement of T25FWT (Timed 25-Foot Walk Test) | 18 weeks
  The difference in the number of patients who achieved an improvement of 20% or more from their baseline T25FWT between those that received 6 weeks of sham rTMS and those that received 6 weeks of rTMS

SECONDARY OUTCOMES:
6MWT (Six minute Walk Test) | 12 weeks
  Patients who achieve an improvement of 30 meters or more in their baseline six Minute Walk Test (6MWT)
MSQoL (Multiple Sclerosis Quality of Life) | 12 weeks
  The change from baseline in MSQoL group mean scores between those that received 6 weeks of sham rTMS and those that received 6 weeks of rTMS

CONTACTS AND LOCATIONS:
Overall Officials: Francois Jacques, Neurologist, Principal Investigator — Clinique Neuro-Outaouais
Locations (1):
- Clinique Neuro-Outaouais, Gatineau, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vickrey BG, Hays RD, Harooni R, Myers LW, Ellison GW. A health-related quality of life measure for multiple sclerosis. Qual Life Res. 1995 Jun;4(3):187-206. doi: 10.1007/BF02260859. PMID 7613530
- [Background] Thompson AJ, Banwell BL, Barkhof F, Carroll WM, Coetzee T, Comi G, Correale J, Fazekas F, Filippi M, Freedman MS, Fujihara K, Galetta SL, Hartung HP, Kappos L, Lublin FD, Marrie RA, Miller AE, Miller DH, Montalban X, Mowry EM, Sorensen PS, Tintore M, Traboulsee AL, Trojano M, Uitdehaag BMJ, Vukusic S, Waubant E, Weinshenker BG, Reingold SC, Cohen JA. Diagnosis of multiple sclerosis: 2017 revisions of the McDonald criteria. Lancet Neurol. 2018 Feb;17(2):162-173. doi: 10.1016/S1474-4422(17)30470-2. Epub 2017 Dec 21. PMID 29275977
- [Background] Schoonheim MM, Meijer KA, Geurts JJ. Network collapse and cognitive impairment in multiple sclerosis. Front Neurol. 2015 Apr 14;6:82. doi: 10.3389/fneur.2015.00082. eCollection 2015. No abstract available. PMID 25926813
- [Background] Rotenberg A, Bae EH, Muller PA, Riviello JJ Jr, Bourgeois BF, Blum AS, Pascual-Leone A. In-session seizures during low-frequency repetitive transcranial magnetic stimulation in patients with epilepsy. Epilepsy Behav. 2009 Oct;16(2):353-5. doi: 10.1016/j.yebeh.2009.08.010. Epub 2009 Sep 10. PMID 19747883
- [Background] Oosterveer DM, van den Berg C, Volker G, Wouda NC, Terluin B, Hoitsma E. Determining the minimal important change of the 6-minute walking test in Multiple Sclerosis patients using a predictive modelling anchor-based method. Mult Scler Relat Disord. 2022 Jan;57:103438. doi: 10.1016/j.msard.2021.103438. Epub 2021 Nov 30. PMID 34871859
- [Background] Joo EY, Han SJ, Chung SH, Cho JW, Seo DW, Hong SB. Antiepileptic effects of low-frequency repetitive transcranial magnetic stimulation by different stimulation durations and locations. Clin Neurophysiol. 2007 Mar;118(3):702-8. doi: 10.1016/j.clinph.2006.11.008. Epub 2007 Jan 16. PMID 17223384
- [Background] Goldman MD, Marrie RA, Cohen JA. Evaluation of the six-minute walk in multiple sclerosis subjects and healthy controls. Mult Scler. 2008 Apr;14(3):383-90. doi: 10.1177/1352458507082607. Epub 2007 Oct 17. PMID 17942508
- [Background] Gandhi OP. Electromagnetic fields: human safety issues. Annu Rev Biomed Eng. 2002;4:211-34. doi: 10.1146/annurev.bioeng.4.020702.153447. Epub 2002 Mar 22. PMID 12117757
- [Background] Barkhof F. The clinico-radiological paradox in multiple sclerosis revisited. Curr Opin Neurol. 2002 Jun;15(3):239-45. doi: 10.1097/00019052-200206000-00003. PMID 12045719
- [Background] Azevedo CJ, Cen SY, Khadka S, Liu S, Kornak J, Shi Y, Zheng L, Hauser SL, Pelletier D. Thalamic atrophy in multiple sclerosis: A magnetic resonance imaging marker of neurodegeneration throughout disease. Ann Neurol. 2018 Feb;83(2):223-234. doi: 10.1002/ana.25150. Epub 2018 Feb 9. PMID 29328531
- [Background] Absinta M, Lassmann H, Trapp BD. Mechanisms underlying progression in multiple sclerosis. Curr Opin Neurol. 2020 Jun;33(3):277-285. doi: 10.1097/WCO.0000000000000818. PMID 32324705
- See also: Clinique Neuro-Outaouais website — https://www.neuro-outaouais.com